CLINICAL TRIAL: NCT02461810
Title: A Prospective, Multicenter, Randomized, Comparative Clinical Study to Compare the Safety and Effectiveness of Two Vertebral Compression Fracture (VCF) Reduction Techniques: the SpineJack® and the KyphX Xpander® Inflatable Bone Tamp
Brief Title: Prospective Comparative Study to Compare Safety and Effectiveness of Two Vertebral Compression Fracture Reduction Techniques
Acronym: SAKOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vexim SA (Industry)
Collaborators: ACES Ing.-GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKOS - EU2014-05
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Spinal Fractures; Vertebral Compression Fractures; Back Injuries; Osteoporosis
MeSH Terms: conditions — Spinal Fractures; Back Injuries; Osteoporosis | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SpineJack® system (Experimental): VCF treatment system Vertebral fracture surgery
  Interventions: Device: Vertebral fracture surgery SpineJack®
- Balloon Kyphoplasty (Active Comparator): VCF treatment system Vertebral fracture surgery
  Interventions: Procedure: Balloon Kyphoplasty

INTERVENTIONS:
Device: Vertebral fracture surgery SpineJack® — Vertebral augmentation for one osteoporotic vertebral compression fracture
  Arms: SpineJack® system
Procedure: Balloon Kyphoplasty
  Arms: Balloon Kyphoplasty

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the SpineJack® with the Kyphx Xpander® Inflatable Bone Tamp and support a non-inferiority finding for the use of SpineJack® VCF treatment system versus Balloon Kyphoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female with at least 50 years of age
2. 1 painful VCF which at least meet all following criteria:

   * Fracture due to diagnosed or presumed underlying osteoporosis
   * VCF between T7 and L3
   * Fracture age <3 months
   * VCF shows loss of height in the anterior, mid or posterior third of the VB from estimated pre-fracture configuration of at least 15% but not more than 40% based on X-Ray at baseline
   * The Index fracture is acute or persistent (not healed), as demonstrated by T2 weighted STIR MRI (or bone scan if patient is contraindicated for MRI)
3. Patient has failed conservative medical therapy, defined as either having a VAS back pain score of ≥50 mm at 6 weeks after initiation of fracture care or a VAS back pain score of ≥70mm at 2 weeks after initiation of fracture care
4. Investigator believes target VB is suitable for SpineJack procedure and Balloon kyphoplasty (e.g., appropriate pedicle diameter) assessed on CT scan pre op
5. Patient has an Oswestry Disability Index (ODI) score of ≥ 30/100
6. Patient is mentally capable and willing to sign a study specific informed consent as documentation of the informed consent process prior to any study procedures
7. The patient is willing and able to comply with all study requirements including follow-up visits and radiographic assessments.

Exclusion Criteria:

1. Target VCF due to underlying or suspected tumor
2. Target VCF due to high-energy trauma
3. Target VCF is diagnosed as an osteonecrotic fracture
4. Segmental kyphosis of target VB of >30°
5. Any prior surgical treatment for a vertebral body compression fracture or other surgical procedure on target VB or adjacent level
6. The patient has uncontrolled diabetes
7. Pre-existing or clinically unstable neurologic deficit
8. The patient has spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level to be treated
9. Any physical exam evidence of myelopathy or radiculopathy
10. The patient has pain based on clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis)
11. Patient not able to walk without assistance prior to fracture
12. Any radiographic evidence of pedicle fracture visible on CT scan pre op
13. Spondylolisthesis >Grade 1 at target VB
14. Any underlying systemic bone disease other than osteoporosis (e.g., osteomalacia, osteogenesis imperfect, Paget's disease, etc.)
15. A medical contraindication to spinal surgery and/or general anesthesia, such as coagulopathy and/or taking warfarin (Coumadin) or other anticoagulant on regular basis for coagulopathy (with a threshold for normal being INR≤1.5, PTT within lab normal range, and platelet count > 100,000)
16. Pain due to any other condition that requires daily narcotic medication
17. Disabling back pain due to causes other than acute fracture
18. History of intolerance or allergic reaction to titanium or acrylic compounds
19. Active systemic or local infection at baseline
20. Body mass index >40
21. Severe cardiopulmonary deficiencies
22. Any other medical illness or condition that, in the investigator's opinion, is likely to impair long-term follow-up (e.g., cancer) or greatly increase the risk of surgery including but not limited to patients with contraindications for general anesthesia (surgeon expertise)
23. Any evidence of alcohol or drug abuse
24. The patient has uncontrolled psychiatric illness or severe dementia
25. The patient is currently on anti-cancer therapy or anti-HIV therapy
26. Patient's life expectancy is less than the study duration or undergoing palliative care
27. Participating in any other investigational study
28. The patient is on long-term steroid therapy (steroid dose ≥ 30 mg /day for > 3 months)
29. The patient is known to be involved in medical litigation including Workmen's Compensation
30. Patient with contraindication for MRI
31. The patient is pregnant or considering getting pregnant during study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-04; Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Study Success | 12 month post-op
  The primary composite endpoint defines a successful subject if the following components are satisfied (safety and effectiveness):
  1. Reduction in VCF fracture-related pain at 12 months from baseline as measured by a 100 mm VAS scale (reduction of pain at 12 months by > 20 mm) AND,
  2. Maintenance or improvement in function at 12 months from baseline as measured by the 100 point Oswestry Disability Index (ODI) AND,
  3. Absence of device-related serious adverse events, defined as device-related adverse events (device migration, recollapse, protrusion) or symptomatic cement extravasation requiring surgical re-intervention or retreatment at the index level, including revision, removal, reoperation, and/or supplemental fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre HONTAS, Director Clinical Affairs, Study Director — Vexim SA
Locations (13):
- France (5):
  - Hôpital Jean Minjoz Service Neurochirurgie, Besançon
  - Centre Hospitalier La Cavale Blanche, Brest
  - CHU La Timone, Marseille
  - Hôpital Nord, Marseille
  - CHU Hôtel Dieu Service Neuro traumatologie, Nantes
- Germany (3):
  - Klinik und Poliklinik fur Orthopädie Universitatsklinikum, Bonn
  - Loretto-Krankenhaus Freiburg, Freiburg im Breisgau
  - Krankenhaus NEUWERK Sankt Augustinus kliniken, Mönchengladbach
- Ospedale SS Trinita ASL8, Cagliari, Italy
- Spain (2):
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valladolid,, Valladolid
- Switzerland (2):
  - HFR Fribourg - Hôpital cantonal, Fribourg
  - Clinique Bois-Cerf, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided